CLINICAL TRIAL: NCT03755011
Title: White Noise to Improve Sleep in the MICU: a Pilot and Feasibility Study
Brief Title: White Noise to Improve Sleep in the Medical Intensive Care Unit (MICU): a Pilot and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000024300
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients exposed to white noise (Experimental): Six patients in the interventional arm will have white noise (through in-room workstations- on-wheels and publicly-available white noise websites) playing overnight at a standardized volume to be determined; pausing will be at nurse, provider, and patient discretion during routine care and conversations with the patients.
  Interventions: Device: white noise
- usual care (Placebo Comparator): Six patients exposed to normal ICU activity noise.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Device: white noise — Patients in the interventional arm will have white noise (through in-room workstations- on-wheels and publicly-available white noise websites) playing overnight at a standardized volume to be determined.
  Arms: patients exposed to white noise
Behavioral: usual care — normal ICU activity noise
  Arms: usual care

SUMMARY:
A feasibility study to evaluate the use of white noise to improve sleeping conditions in an ICU setting.

DETAILED DESCRIPTION:
The ICU is full of alarms and critically ill patients, so it is no surprise that sleep is very much fragmented and poor in this setting, as documented in numerous studies. White noise is a simple intervention that has been shown to improve sleep, including in the ICU setting. The aim is to conduct a pilot trial evaluating the feasibility of providing white noise to patients in the ICU at night to help improve sleep. The plan to measure feasibility metrics including patient acceptance, patient tolerance, and intervention fidelity; also to seek feedback from patients, nurses, and providers. Secondly is to evaluate the benefits of providing white noise at night in the ICU on sleep as measured by actigraphy and Richards-Campbell Sleep Questionnaires and total room sound.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18yo admitted to MICU with expected stay of at least two nights after enrollment

Exclusion Criteria:

* Excluding intubated patients (so communication can be better) and patients on high-flow nasal cannula (which is already high background noise).
* Patients who are on therapeutic hypothermia or are on comfort measures only will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Intervention fidelity: percent of intervention time during which white noise is actually delivered | 48 hours
  percent of intervention time during which white noise is actually delivered

SECONDARY OUTCOMES:
Sound Levels | 48 hours
  Room dBA and dBC-weighted sound levels will be measured in the rooms as well by HD600 sound meters (Extech Instruments) every 10 seconds throughout the night shift; sound meters will be placed on the wall behind and 10" above the head of the bed (set when head of bed is at 30 degrees).
Sleep Questionnaire: Sleep Questionnaire. Patients will be surveyed after Study Night 1 and Study Night 2 with Richards- Campbell Sleep Questionnaires. | 48 hours
  Sleep Questionnaire. Patients will be surveyed after Study Night 1 and Study Night 2 with Richards- Campbell Sleep Questionnaires. Scores will be graded on a scale of 0-100, as measured in mm on the visual scale; 100 representing a more positive sleep experience.
Actigraphic rest-activity :Patients will wear Actiwatch Spectrum devices to measure rest-activity patterns. Sleep will be identified using Actiwatch Software as provided by the manufacture. | 48 hours
  Patients will wear Actiwatch Spectrum devices to measure rest-activity patterns. Sleep will be identified using Actiwatch Software as provided by the manufacture.
Patient tolerance: percent of days that patients agree to continue white noise | 48 hours
  percent of days that patients agree to continue white noise
Patient acceptance: percent of patients or surrogates who agree to receive white noise at night | 48 hours
  percent of patients or surrogates who agree to receive white noise at night

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Gao, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States